CLINICAL TRIAL: NCT07326410
Title: Prevalence of Cerebral Large Vessel Occlusion Among Acute Ischemic Stroke Patients in Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Tarek Aly Sayed, Resident of neurology, Assiut University
Other Study IDs: Prevalence of Cerebral LVO
Record Dates: First submitted 2025-12-08; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
Keywords: Prevalence of cerebral Large Vessel Occlusion among acute ischemic stroke patients
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence of Large Vessel Occlusion among acute ischemic stroke patients in Assiut University hospitals

1. Study Objectives

   Primary Objective:

   - To determine the prevalence of LVO among acute ischemic stroke (AIS) patients presenting to Assiut University hospitals

   Secondary Objectives:
   * To describe clinical and radiological characteristics of LVO patients.
   * To assess factors associated with LVO (age, sex, stroke severity, comorbidities).
2. Study Design

   * Type: single center, prospective observational cross-sectional study
   * Duration: 12-month recruitment period
   * Setting: Assiut university hospitals, stroke unit.
3. Study Population

Inclusion Criteria:

* Adults (≥18 years)
* Diagnosed with acute ischemic stroke within 24 hours of symptom onset
* Underwent vascular imaging (CTA or MRA) on admission

Exclusion Criteria:

* Hemorrhagic stroke
* Stroke mimics
* Incomplete imaging data 4. Definitions

Large Vessel Occlusion (LVO) defined as occlusion in:

* Intracranial ICA
* M1 or proximal M2 segments of MCA
* Basilar artery ± Optional: A1 6. Data Collection

Clinical Data:

* Demographics (age, sex)
* Risk factors (HTN, DM, AF, CAD, smoking)
* NIHSS on admission and discharge mRS on admission and discharge
* Onset-to-door time
* Imaging modality used

Imaging Data:

* Site of occlusion
* ASPECTS (optional)
* Collateral status (optional if available)

Hospital Data:

* Facility type (public vs private)
* Door-to-CT and door-to-CTA times 8. Analysis Plan
* Primary: Prevalence of LVO = Number of LVO cases / Total AIS patients with vascular imaging
* Subgroup analysis: By age group, sex, region, NIHSS
* Secondary: Logistic regression to identify predictors of LVO

DETAILED DESCRIPTION:
Prevalence of Large Vessel Occlusion among acute ischemic stroke patients in Assiut University hospitals

1. Study Objectives

   Primary Objective:

   - To determine the prevalence of LVO among acute ischemic stroke (AIS) patients presenting to Assiut University hospitals

   Secondary Objectives:
   * To describe clinical and radiological characteristics of LVO patients.
   * To assess factors associated with LVO (age, sex, stroke severity, comorbidities).
2. Study Design

   * Type: single center, prospective observational cross-sectional study
   * Duration: 12-month recruitment period
   * Setting: Assiut university hospitals, stroke unit.
3. Study Population

Inclusion Criteria:

* Adults (≥18 years)
* Diagnosed with acute ischemic stroke within 24 hours of symptom onset
* Underwent vascular imaging (CTA or MRA) on admission

Exclusion Criteria:

* Hemorrhagic stroke
* Stroke mimics
* Incomplete imaging data 4. Definitions

Large Vessel Occlusion (LVO) defined as occlusion in:

* Intracranial ICA
* M1 or proximal M2 segments of MCA
* Basilar artery ± Optional: A1 6. Data Collection

Clinical Data:

* Demographics (age, sex)
* Risk factors (HTN, DM, AF, CAD, smoking)
* NIHSS on admission and discharge mRS on admission and discharge
* Onset-to-door time
* Imaging modality used

Imaging Data:

* Site of occlusion
* ASPECTS (optional)
* Collateral status (optional if available)

Hospital Data:

* Facility type (public vs private)
* Door-to-CT and door-to-CTA times 8. Analysis Plan
* Primary: Prevalence of LVO = Number of LVO cases / Total AIS patients with vascular imaging
* Subgroup analysis: By age group, sex, region, NIHSS
* Secondary: Logistic regression to identify predictors of LVO

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Diagnosed with acute ischemic stroke within 24 hours of symptom onset
* Underwent vascular imaging (CTA or MRA) on admission

Exclusion Criteria:

* Hemorrhagic stroke
* Stroke mimics
* Incomplete imaging data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Large Vessel Occlusion (LVO) defined as occlusion in:
  * Intracranial ICA
  * M1 or proximal M2 segments of MCA
  * Basilar artery ± Optional: A1
  Clinical Data:
  * Demographics (age, sex)
  * Risk factors (HTN, DM, AF, CAD, smoking)
  * NIHSS on admission and discharge mRS on admission and discharge
  * Onset-to-door time
  * Imaging modality used
  Imaging Data:
  * Site of occlusion
  * ASPECTS (optional)
  * Collateral status (optional if available)
  Hospital Data:
  * Facility type (public vs private)
  * Door-to-CT and door-to-CTA times
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
To determine the prevalence of LVO among acute ischemic stroke (AIS) patients presenting to Assiut University hospitals | 12 months
  Prevalence of LVO = Number of LVO cases / Total AIS patients with vascular imaging

SECONDARY OUTCOMES:
-To describe clinical and radiological characteristics of LVO patients. - To assess factors associated with LVO (age, sex, stroke severity, comorbidities). | 12 months
  Subgroup analysis: By age group, sex, region, NIHSS

IPD SHARING:
Plan to Share IPD: No
Financial issues

REFERENCES:
- See also: Prevalence of cerebral Large Vessel Occlusion among acute ischemic stroke — https://pubmed.ncbi.nlm.nih.gov/30415226/